CLINICAL TRIAL: NCT01330784
Title: Assessment of the Therapeutic Utility of hMG-HP Within a Protocol of Controlled Ovarian Hyperstimulation in IVF in Normoresponders Women Undergoing Downregulation With GnRH Antagonist
Brief Title: Assessment of the Therapeutic Utility of hMG-HP
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring SAU (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Other Study IDs: FER-GON-2004-02
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Sterility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hMG-HP: Patients with a condition
  Interventions: Drug: hMG-HP

INTERVENTIONS:
Drug: hMG-HP

SUMMARY:
To assess the effectiveness of a protocol of ovarian hyperstimulation with urinary gonadotrophins, to achieve clinical pregnancy in females undergoing IVF.

Study hypothesis: to assess the effectiveness of a protocol of urinary gonadotrophins

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-38 years
* Body mass index (BMI) between 18 and 30
* Women classified as normogonadotrophin patients. Not more than 3 previous cycles of ART (assisted reproductive technology)
* Testosterona, FSH (follicle-stimulating hormone) LH (luteinizing hormone) and Prolactin serum levels during the early folicular phase (days 2-4 of the cycle) within the laboratory normal range
* No administration of clomiphen citrate or gonadotropins during the month prior to the start of the study

Exclusion Criteria:

* Failure in previous cycles of assisted reproduction IVF/ICSI (in-vitro fertilisation/intracytoplasmic sperm injection)
* Seminal samples not apt for IVF-ICSI (according to the criteria of each center). Evidence of significant bacterial infection in the seminogram of the couple in the preceding 6 months
* Data suggestive of possible ovarian failure
* Antecedents of severe ovarian hyperstimulation syndrome (OHSS)
* Important systemic disease
* Pregnancy or contraindication to pregnancy

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females affected by sterility able to undergo IVF
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 30 days

SECONDARY OUTCOMES:
Biochemical pregnancy rate | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Investigational site, Valencia, Valencia, Spain